CLINICAL TRIAL: NCT04136483
Title: Cognitive-behavioral Therapy for Insomnia in Adolescent Psychiatry: a Clinical Pilot Study
Brief Title: Cognitive-behavioral Therapy for Insomnia in Adolescent Psychiatry
Acronym: 2012/871-31/1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm University (Other); Child and Adolescent Psychiatry, Stockholm (Industry); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Lekander, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-871-31-1
Record Dates: First submitted 2019-09-03; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT-I (Experimental)
  Interventions: Behavioral: CBT-I

INTERVENTIONS:
Behavioral: CBT-I — The theoretical framework is cognitive-behavioral therapy that includes sleep education, sleep hygiene, sleep restriction, stimulus control, cognitive interventions and relaxation. The intervention has been adapted to adolescents by reducing the amount of psychoeducational information and the interventions related to changing cognitions. It involves six weekly face-to-face individual sessions with a therapist, supported by a participant workbook that contains information, work- sheets, and at-home tasks. Clinical psychologists or graduate clinical psychologists in training delivered the intervention sessions under supervision by the first author. Parents/care-givers were given information about the components, but did not take active part of the intervention.

SUMMARY:
The study is a clinical pilot study that examine the preliminary effect of cognitive-behavioral therapy for insomnia (CBT-I) in adolescents with comorbid psychiatric disorders. Participants (n=25) are recruited from three psychiatric clinics (n=19) and one pediatric pain clinic (n=6). After diagnostic assessment, participants that fulfil inclusion criteria are offered the CBT-I intervention. Pre-post and 3-months follow-up assessments include subjective measures of insomnia symptom severity, sleep parameters (collected through sleep-wake diaries), symptoms of depression and anxiety and daytime functioning.

ELIGIBILITY:
Inclusion Criteria:

* be between 13-17 years old
* meet criteria for insomnia disorder (primary or secondary insomnia) according to DSM-IV-TR
* have insomnia symptoms at a clinical level, as defined as more than 10 points on the ISI-a
* adequate Swedish language skills

Exclusion Criteria:

* severe psychiatric disorder that is contraindicative of the treatment (i.e., bipolar disorder, psychotic disorder)
* autistic disorder
* severe suicidality (defined as ≥17 points on MINI-kid suicide subscale)
* alcohol or drug dependence
* psychotropic medication
* previous (> 5 sessions) or ongoing CBT-treatment for insomnia

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Insomnia Severity Index- adolescent version (ISI-a) | 6 weeks and 3 months
  The Insomnia Severity Index, ISI -adolescent version18 was used before, after at three months follow-up to measure insomnia symptom severity. ISI-a is an adaptation to adolescents of the Insomnia Severity Index32,36. ISI-a is a seven-item measure that yields a quantitative index of sleep impairment and treatment outcome. Total scores range from 0 to 28, with higher scores indicating greater perceived insomnia severity.

SECONDARY OUTCOMES:
Sleep Onset Latency (SOL) | Baseline, 6 weeks and 3 months
  Subjective sleep onset latency was measured using a sleep-wake diary (SWD) before, after and at three-months follow-up. Participants filled in the SWD during seven consecutive days/nights at all time points.
Wake after sleep onset (WASO) | Baseline, 6 weeks and 3 months
  Subjective wake after sleep onset was measured using a sleep-wake diary (SWD) before, after and at three-months follow-up. Participants filled in the SWD during seven consecutive days/nights at all time points.
Total Sleep Time (TST) | Baseline, 6 weeks and 3 months
  Subjective total sleep time was measured using a sleep-wake diary (SWD) before, after and at three-months follow-up. Participants filled in the SWD during seven consecutive days/nights at all time points.
Sleep Efficiency (SE) | Baseline, 6 weeks and 3 months
  Subjective sleep efficiency was measured using a sleep-wake diary (SWD) before, after and at three-months follow-up. Participants filled in the SWD during seven consecutive days/nights at all time points.
Spences' Children Anxiety Scale (SCAS) | Baseline, 6 weeks and 3 months
  Spences Children's Anxiety Scale - SCAS 37 was used before, after and at three months follow-up to measure level of anxiety symptoms. SCAS is a child self-report measure of anxiety related psychopathology, measuring five domains of anxiety: generalized anxiety, panic anxiety, separation anxiety, social anxiety and obsessive-compulsive anxiety.Scores range from 0 to 114 and higher scores indicate more severe symptoms of anxiety.
Center for Epidemiological Studies Depression Scale for Children (CES-DC) | Baseline, 6 weeks and 3 months
  Center for Epidemiological Studies Depression Scale for Children (CES-DC)38 was used before, after and at three months follow-up to measure depressive symptoms. CES-DC is a 20-item self-report depression inventory.Scores range from 0 to 60, with higher scores indicating more severe depressive symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Mats Lekander, Professor, Principal Investigator — Karolinska Institutet